CLINICAL TRIAL: NCT00505882
Title: The Pilot Study:Efficacy of Pramlintide on Prevention of Weight Gain Early Onset of Type 1 Diabetes
Brief Title: Efficacy of Pramlintide on Prevention of Weight Gain Early Onset of Type 1 Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Philip Raskin, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 032007-054
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Pramlintide; Weight gain; Intensive insulin therapy; Beta cell
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Weight Gain | interventions — pramlintide; Insulin Glargine; Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Active Comparator)
  Interventions: Drug: Glargine; Drug: Lispro; Drug: Aspart
- Pramlintide (Experimental)
  Interventions: Drug: Pramlintide; Drug: Glargine; Drug: Lispro; Drug: Aspart

INTERVENTIONS:
Drug: Pramlintide — Pramlintide will be started at 15 mcg (2.5 units) subcutaneously immediately prior to major meals and it will be increased by 15mcg every 3 days as tolerated (i.e. nausea, vomiting, upset stomach) to a maximum dose of 60 mcg (10 units) before meals. If significant nausea persists at 45 or 60 mcg level, the dose should be decreased to 30 mcg (5 units) before meals. If the 30 mcg dose is not tolerated, investigator will evaluate for possibility of withdrawing the pramlintide. The dose of preprandial short acting insulin (eg: Novolog/Humalog) will be reduced by 30 to 50% at the start of pramlintide 15 mcg (2.5 units) and then will be adjusted every time the dose of pramlintide is increased by 15 mcg (2.5 units) as needed based on blood glucose readings.
  Other Names: Symlin
  Arms: Pramlintide
Drug: Glargine
Drug: Lispro
Drug: Aspart

SUMMARY:
In this pilot study we are evaluating the efficacy of pramlintide on preventing weight gain among early onset type 1 diabetes. We are also evaluating the safety and the effects of treatment with pramlintide on early diagnosed type 1 diabetic subjects, especially among pediatric subjects.

DETAILED DESCRIPTION:
The autoimmune process along with a strong genetic-mediated destruction and dysfunction of pancreatic β-cells are the main pathogeneses of type 1 diabetes. These processes cause absolute and relative insulin and amylin deficiencies. For the last decades, insulin therapy has been the primary therapy for type 1 diabetes.

Amylin is a 37 amino acid peptide hormone co-secreted with insulin mostly by the pancreatic β cells in response to meals. Amylin has several known effects including suppression of postprandial glucagon secretion, regulation of gastric emptying, and reduction of food intake. Pramlintide is an amylin analog recently approved by the Food and Drug Administration (FDA) to be given at meal time as an adjunct to insulin therapy in patients with type 1 or type 2 diabetes who have failed to achieve desired glucose control despite optimal insulin therapy or insulin therapy with or without a sulfonylurea agent and/or metformin. Several clinical trials showed that meal time amylin replacement with pramlintide along with insulin therapy improved post-prandial hyperglucagonemia, and reduced post-prandial glucose excursion. A recent randomized control trial showed that pramlintaide reduced weight by up to 2kg in both type 1 and type 2 diabetes.

The Diabetes Control and Complications Trial (DCCT) demonstrated that intensive diabetes therapy delays the onset and progression of microvascular disease such as retinopathy, nephropathy and neuropathy. The DCCT also showed that the prevalence of obesity, defined as a body mass index (BMI) ≥ 27.8 kg/m2 for men and ≥ 27.3 kg/m2 for women, was 33.1% in the intensive treatment group compared with 19.1% in the conventional treatment group. Intensively treated patients gained an average of 4.75 kg more than conventionally treated patients (P < 0.0001). Weight gain was most rapid during the first year of therapy. Several mechanisms have been proposed to explain the weight gain associated with insulin therapy. These include decreased glycosuria due to improved glycemic control, the direct lipogenic effects of insulin on adipose tissue, and increased food intake due to recurrent mild hypoglycemia.

Obesity, especially in type 2 diabetes, is associated with the accumulation of triglyceride in muscle as well as in the liver. These are thought to cause insulin resistance and diabetic metabolic complications. Sub-analysis of the DCCT showed that in the intensive treatment group, higher weight gain correlated with a higher waist to hip ratio as well as higher LDL and lower HDL levels similar to what is seen in the metabolic syndrome. An association between weight gain due to intensive insulin therapy in type 1 diabetes and the risk of coronary artery disease has yet to be determined. However, the DCCT showed some reduction in cardiovascular risk factors among the intensive treatment group as well as reduction in cardiovascular events. The DCCT did not evaluate cardiovascular risk based on degree of obesity within the intensive insulin treatment group.

The DCCT has shown that the intensive insulin therapy group maintained a higher stimulated C-peptide level than the conventional group. Preserving β cell function, even modest levels of activity can be advantage in preventing hypoglycemic episodes and also reducing the incidence of retinopathy and nephropathy. No study to date has been designed to analyze the effect of pramlintide treatment on the preservation of β cell function in newly diagnosed type 1 diabetic subjects.

This pilot study will evaluate the effect of pramlintide on the prevention of weight gain and its effects on beta cell function among early onset type 1 diabetes patients. Early onset is defined as those who are diagnosed with type 1 diabetes six to twelve months prior to entry in this study.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 40 years old
* Type 1 diabetes
* Fasting C-peptide ≤ 1.0 ng/ml
* Early diagnosed type 1 diabetes. (<6 months since diagnosis of type 1 diabetes.)
* HbA1c greater than 7.0 %
* Male, or If female, is nonlactating and has a negative pregnancy test (human chorionic gonadotropin, beta subunit [βhCG]) at Visit 1 (screening).

Exclusion Criteria:

* Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

  * Hepatic disease
  * Gastrointestinal disease
  * Haematologic disorder
  * Cardiovascular disorder
  * Organ transplantation
  * Hemochromatosis
  * HIV, HBV, or HCV infection
* Abuses drugs or alcohol or has a history of abuse
* Eating disorder
* Has donated blood within 60 days
* Has had major surgery or a blood transfusion within 2 months
* Usage of medications that affect weight changes
* Use of medications that affect gastrointestinal motility
* Usage of medications that affect glucose/insulin metabolism
* Received any study medication or has participated in any type of clinical trial within 30 days prior to screening.
* Has known allergies or hypersensitivity to any component of study treatment.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The change in weight (kg) will be compared between as well as within the placebo and the pramlintide treatment group from baseline to the end of the study. | 6 months

SECONDARY OUTCOMES:
mixed meal tolerance test-the C-peptide area under the curve The HOMA R and McAuley's index HbA1c The event rate of severe hypoglycemia Waist circumference Cardio C-reactive protein level DQOL Safety parameter | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Raskin, M.D., Principal Investigator — UT Southwestern at Dallas
Locations (1):
- UT Southwestern at Dallas, Dallas, Texas, United States